CLINICAL TRIAL: NCT05154448
Title: High-Intensity Focused Ultrasound Ablation With the Neurolyser XR Device for the Treatment of Chronic Low Back Pain: a Prospective Randomized Double-Blind Sham-Controlled Multicenter Study
Brief Title: Double Arm Pivotal Study to Evaluate the Neurolyser XR for the Treatment of Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FUSMobile Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LBP003
Record Dates: First submitted 2021-11-16; First posted 2021-12-13 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2023-10

CONDITIONS: Facet Syndrome of Lumbar Spine
Keywords: chronic low back pain; zygapophyseal joint syndrome; Facet syndrome

STUDY DESIGN:
Intervention Model Description: Double arm randomized study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The sham procedure would be done using the same system and setup. Randomization would be done using an EDC system and no person at the room would know if the procedure is a treat or sham procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Thermal ablation of the medial nerve branch using High Intensity Focused Ultrasound (Experimental): Non-Invasive Thermal Ablation of the Medial Branch Nerves using the Neurolyser XR High Intensity Focused Ultrasound device
  Interventions: Device: Non-Invasive Thermal Ablation of the Medial Branch Nerves (Neurolyser XR)
- Sham treatment (Sham Comparator): The procedure would be done in an identical manner to the NeurolyserXR treatment without any person in the procedure room knowing that this is a sham procedure.
  The only difference is that the acoustic energy would not be output from the system during a sham procedure.
  Interventions: Other: Sham procedure

INTERVENTIONS:
Device: Non-Invasive Thermal Ablation of the Medial Branch Nerves (Neurolyser XR) — Thermal ablation of the medial nerve branch using High Intensity Focused Ultrasound
  Arms: Thermal ablation of the medial nerve branch using High Intensity Focused Ultrasound
Other: Sham procedure — Sham procedure done in an identical manner to the treatment arm, but without deploying acoustical energy
  Arms: Sham treatment

SUMMARY:
Double arm pivotal study to evaluate the Neurolyser XR as a non-invasive treatment of axial chronic low back pain

DETAILED DESCRIPTION:
Study design: Prospective, Double Arm Timeline: Twelve months enrollment period and 6 months follow-up period. Sites: The study will be conducted at 10 sites in the USA Study population: 80 adult subjects diagnosed with facet related low back pain with an additional 10 roll in subjects.

Arms: 40 patients would be treated by the NeurolyserXR and 40 would get a sham treatment Crossover: blinded crossover between the two arms could be done between 1 and 3 months Primary study objective: Safety and efficacy of the Neurolyser XR for the treatment of chronic low back pain secondary to zygapophyseal joint syndrome.

Safety is measured by the incidence and severity of treatment related adverse events.

Efficacy is measured by pain numerical rating scale

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 to 85 years old, legally able and willing to participate in the study and all follow-up visits
2. Able and willing to complete the research questionnaires and to communicate with investigator and research team
3. Individual with current bilateral or unilateral low back pain of > 6 months duration
4. Individual whose back pain is alleviated by recumbency or comfortable sitting position
5. Individual presenting with a) a positive (>80% pain relief) to a previous, double, lumbar medial branch block (within the last 12 months) and/or b) with a positive (>70% pain relief lasting more than 6 months) to the most recent lumbar facet thermal radiofrequency denervation
6. Average low back pain score of 6 or higher in the last month (on 0-10 scale) with activity

Exclusion Criteria:

1. Individuals who are pregnant or breastfeeding
2. Individuals younger than 50 or older than 85 years
3. BMI greater than 40, or individuals with at least one of the planned targets outside the Neurolyser XR treatment envelope as seen on treatment day on a lateral X-ray scan taken before the treatment.
4. Individuals presenting with neurological deficits (including lumbosacral radiculopathy but not solitary radicular pain)
5. Individuals with history of lumbar or lumbosacral spine surgery
6. Individuals who have had lumbar radiofrequency neurotomy in the past 6 months
7. Individuals with history of lumbar spine pathology that may increase procedural risk and/or influence symptoms and/or generate unrelated adverse event (per investigator's discretion)
8. Individuals presenting with any severe medical condition preventing them from participation (per investigator's discretion) (Example: inability to lay prone)
9. Individuals with extensive scarring of the skin and tissue overlying the treatment area
10. Individuals enrolled in or planned to be enrolled in another clinical trial during the duration of this research project
11. Any Individuals with an uncontrolled coagulopathy
12. Individuals with known osteoporosis with absolute risk of spinal fracture of > 10% over 10 years
13. Any Individuals with a history of malignant disease in the past five years or any individuals with clinical history suggestive of new/previously unknown malignancy and pathological pain who require further work up or is currently undergoing work up
14. Individuals with rheumatologic diseases causing spine pain that are currently receiving active treatment including steroids, disease modifying drugs, biological agents or immunosuppressants
15. Individuals known for concomitant psychiatric disorders, excluding compensated mood disorders
16. Individuals with first-degree family member already enrolled in this study
17. Individual who is scheduled for any interventional/surgical procedure within 6 months from the treatment date excluding trivial surgeries (e.g., cataract, carpal tunnel release)
18. Individuals diagnosed with co-morbid multifocal chronic pain (e.g. fibromyalgia, generalized osteoarthritis)
19. Individuals with other chronic pain that is 2 or more points higher on the NRS score than the participants low back pain
20. Individuals who have had a steroid injection within the last 2 months from date of enrollment at the location of the planned treatment
21. Any individuals with clinical or radiographic evidence of dynamic instability of the lumbar spine

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
NRS | Base line, 2 days 1, 2 & 4 weeks, 3 & 6 months after procedure
  Change in average pain score as measured by a numeric rating scale from 0 (no pain) to 10, worst possible pain
Procedure and Device Safety up to six months post procedure | 6 months after procedure
  Safety will be measured by the incidence and severity of treatment related adverse events

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | Time Frame: Base line, 1, & 4 weeks, 3 & 6 months after procedure
  Low Back Pain Questionnaire (Range: 0% to 100%)
Patient Global Impression of Change (PGIC) | Time Frame: Base line, 1, & 4 weeks, 3 & 6 months after procedure
  Patient Global Impression of Change (Range: 1 to 7)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Stamford Hospital, Stamford, Connecticut
  - Mayo University Jacksonville, Jacksonville, Florida
  - Univ of Miami Rehabilitation Medicine, Miami, Florida
  - Emory, Atlanta, Georgia
  - The Physicians Spine and Rehabilitation Specialist of GA, Atlanta, Georgia
  - Charlie Norwood VA Medical Center, Augusta, Georgia
  - Ainsworth Institute of Pain Management, New York, New York
  - Center for Clinical Research, Winston-Salem, North Carolina
  - University of Virginia Pain Management Center, Charlottesville, Virginia
  - Gershon Pain Specialists, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No